CLINICAL TRIAL: NCT05497544
Title: A Randomized Controlled Trial to Evaluate the Impact of Oncologists 'Exercise Recommendation on the Exercise Levels in Lung Cancer Patients
Brief Title: ORE - 30 Seconds (Oncologists Recommend Exercise in 30 Secs)
Acronym: ORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alice Avancini, Co-investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 26622
Record Dates: First submitted 2022-08-06; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise recommendation group (Experimental)
  Interventions: Behavioral: Exercise recommendation group
- Exercise recommendation plus guidebook group (Experimental)
  Interventions: Behavioral: Exercise recommendation plus guidebook group
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Exercise recommendation group — A verbal exercise recommendation will be provided. This recommendation will be reported also in the hospital resignation letter.
  Arms: Exercise recommendation group
Behavioral: Exercise recommendation plus guidebook group — This group will receive the exercise (verbal and written) recommendation. Additionally, the oncologist hand the patient a guidebook about exercise, specifically designed for cancer patients.
  Arms: Exercise recommendation plus guidebook group

SUMMARY:
The O.R.E. - 30 seconds (Oncologists Recommend Exercise in 30 secs) trial aims to test the impact of oncologist recommendations on physical activity level, in patients with lung cancer.

DETAILED DESCRIPTION:
Lung malignancy still remains the leading cause of cancer incidence and mortality worldwide. Despite the improvement in terms of innovative treatments, lung cancer and related therapies continue to be associated with severe physical, psychological, and social side effects.

In recent years, several studies have investigated the potential role of physical activity (PA) and exercise (EX) as supportive therapy following a lung cancer diagnosis. Several randomized controlled studies provided evidence that EX is safe for lung cancer patients and may enhance several physiologic and psychologic outcomes. During the preoperative period, EX has demonstrated to increase cardiorespiratory fitness (CRF), and muscular strength, to reduce postoperative complications and length of hospital stay. Following surgery and/or during medical treatments, EX has shown to have a potent modulator effect, able to increase the health-related fitness capacities (especially CRF, muscular strength, and body composition), manage some treatment side effects, such as cancer-related fatigue, sleep disorder and anxiety/depression symptoms. In lung cancer settings, health-related fitness capacities, especially CRF, muscular strength and body composition, are resulted to be prognostic factors. For example, Jones et al. prospectively found that each 50 meters improvement in six minutes walking test (for assessing CRF) was associated with a reduction of 13% in the risk of death in patients with metastatic non-small cell lung cancer. Moreover, some preliminary observational data suggest that higher postdiagnosis PA is associated with lower recurrence, and specific and all-cause mortality in breast, colon, and prostate cancers. American Cancer Society and the American College of Sports Medicine recommend that cancer patients should achieve at least 90 min of moderate-intensity aerobic physical activity each week, with strength and flexibility exercises at least two times per week.

Though the EX benefits are remarkable, most lung cancer patients result insufficiently active. Physician counseling has a positive impact on physical activity levels in sedentary adults, and even in the oncological setting can be a crucial key to engaging or improving PA or EX. Lung cancer patients reported that they prefer to receive PA information primarily from oncologists, and this counseling seems effective in improving PA levels. A randomized controlled trial indicated that 30-second oncologist counseling has a modest effect on PA behavior in breast cancer patients. In particular, at five weeks post-consultation, patients that received EX recommendation reported 3.4 metabolic equivalents of the task (MET)-hour of total EX per week (approximately 30 minutes of moderate-intensity) more compared to the usual care group.

To date, limited data support the favorable role of oncologist recommendation, with no research focusing on lung cancer settings. To bridge this gap, we propose the O.R.E. - 30 seconds (Oncologists Recommend Exercise in 30 secs) trial to test the impact of oncologist recommendation on physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of lung cancer (from 0 to 24 months since diagnosis;
* Stage I-IV;
* Age ≥ 18 years;
* ECOG (performance status) ≤ 1;
* Written informed consent signed.

Exclusion Criteria:

* Obvious significant physical or psychological disabilities (e.g., wheelchair, severe anxiety);
* Not able to speak, read or write in Italian;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Exercise level | Change from baseline to 4 weeks
  Exercise level will be evaluated with Godin's Shepard Leisure Time Exercise Questionnaire (0-700)

SECONDARY OUTCOMES:
Sedentary behavior | Change from baseline to 4 weeks
  Sedentary behavior will be evaluated with the sedentary Behavior Questionnaire (0-500)
Quality of life | Change from baseline to 4 weeks
  Quality of life will be evaluated with the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (0-100)

OTHER OUTCOMES:
Overall survival | Change from baseline to12 months
  Overall survival will be assessed through death from any cause.
Progression free survival | Change from baseline to 12 months
  Progression free survival will be assessed through tumor progression or death from any cause
Treatment-related side effects | Change from baseline to 12 months
  Treatment-related side effects will be assessed using the Common Terminology Criteria for Adverse Events
Exercise level | Change from baseline to 8 weeks
  Exercise level will be evaluated with Godin's Shepard Leisure Time Exercise Questionnaire (0-700)
Sedentary behavior | Change from baseline to 8 weeks
  Sedentary behavior will be evaluated with the sedentary Behavior Questionnaire (0-500)
Quality of life | Change from baseline to 8 weeks
  Quality of life will be evaluated with the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona, Verona, Italy